CLINICAL TRIAL: NCT04926129
Title: Natural History of the Progression of X-Linked Retinitis Pigmentosa
Acronym: XOLARIS
Status: Completed | Type: Observational
Sponsor: NightstaRx Ltd, a Biogen Company (Other)
Responsible Party: Sponsor
Organization: Biogen (Industry)
Other Study IDs: 274RP001; NSR-XLRP-OS1 (Other: NightstaRx Ltd, a Biogen Company)
Record Dates: First submitted 2019-07-30; First posted 2021-06-14 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: X-Linked Retinitis Pigmentosa
Keywords: RP GTPase regulator (RPGR); Degenerative retinal disease; XLRP; Natural history; Rare disease
MeSH Terms: conditions — Rare Diseases | interventions — Cotoretigene Toliparvovec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subgroup 1: Participant's eye with Early Treatment Diabetic Retinopathy Study (ETDRS) best-corrected visual acuity (BCVA) ≥74 letters (Equivalent to: Snellen 6/9 or 20/32; decimal 0.63; Logarithm of the minimum angle of resolution [LogMAR] 0.2) will be enrolled.
  Interventions: Other: Other: Assessments
- Subgroup 2: Participant's eye with ETDRS BCVA 34-73 letters, inclusive (Equivalent to: Snellen 6/12 - 6/60 or 20/40 - 20/200; decimal 0.5 - 0.1; LogMAR 0.3-1.0) will be enrolled.
  Interventions: Other: Other: Assessments

INTERVENTIONS:
Other: Other: Assessments — Administered as specified in the treatment arm.
  Other Names: BIIB112

SUMMARY:
The objective of the study is to gain a better understanding of disease progression over time in participants with X-linked retinitis pigmentosa (XLRP).

DETAILED DESCRIPTION:
This study was previously posted by NightstaRx Ltd. In October, 2020, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have documentation of a pathogenic mutation in the retinitis pigmentosa GTPase regulator (RPGR) gene.
2. Are willing and able to undergo ophthalmic examinations, as required by protocol, for up to 24 months
3. Have an ETDRS BCVA in at least 1 eye of ≥34 letters (Equivalent to Snellen ≥ 6/60 or 20/200; decimal 0.1; LogMAR 1.0).
4. Mean retinal sensitivity in the eligible eye as assessed by microperimetry:

   * Males with a mean retinal sensitivity of 68 loci ranging from ≥0.1 decibels (dB) and ≤20 dB.
   * Females with a mean retinal sensitivity of 68 loci ranging from ≥0.1 dB and ≤25 dB.
5. If female, have symptomatic disease with impairment of visual function.

Key Exclusion Criteria:

1. Have a history of amblyopia in the eligible eye.
2. Have any other significant ocular or non-ocular disease/disorder which, in the opinion of the investigator, may put the participant at risk because of participation in the study, may influence the results of the study, may influence the participant's ability to perform study diagnostic tests, or impact the participant's ability to participate in the study. This includes clinically significant cataracts.
3. Have participated in another research study involving an investigational medicinal product in the past 12 weeks or received a gene/cell-based therapy at any time previously (including but not limited to Intelligent Implant System implantation, ciliary neurotrophic factor therapy, nerve growth factor therapy).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 201 participants with X-linked Retinitis Pigmentosa (XLRP).
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) | Up to Month 24
  BCVA will be assessed for both eyes using the ETDRS visual acuity (VA) chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. BCVA is to be reported as number of letters read correctly by the participant.
Change from Baseline in Retinal Sensitivity Assessed with Microperimetry | Up to Month 24
  Macular analyser integrity assessment (MAIA) microperimetry will be conducted for both eyes to assess changes in retinal sensitivity within the macula.

SECONDARY OUTCOMES:
Change from Baseline in Contrast Sensitivity | Up to Month 24
  Change from baseline in contrast sensitivity in the study eye is measured using a Pelli Robson contrast sensitivity chart at 1 meter. The contrast sensitivity chart contains letters that are darkest at the top and then get progressively lighter. Scores range from 0 to 48 and are based on the number of letters read correctly. A negative change from baseline indicates a worsening in contrast sensitivity and a positive change from baseline indicates an improvement.
Change from Baseline in Low Luminance Visual Acuity (LLVA) | Up to Month 24
  LLVA is measured by placing a 2.0-log-unit neutral density filter over the front of each eye and having the participant read the normally illuminated ETDRS chart. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. LLVA is to be reported as number of letters read correctly by the participant.
Change from Baseline in 25-item Visual Function Questionnaire (VFQ-25) Score | Up to Month 24
  VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. In this format scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score.
Change from Baseline in Retinitis Pigmentosa (RP)-Specific Patient-Reported Outcome (PRO) Questionnaire | Up to Month 24
Change from Baseline in EuroQol-5 Dimension 5-level (EQ-5D-5L) | Up to Month 24
  The widely validated EQ-5D includes 2 components, the EQ-5D descriptive system and the EQ VAS. The EQ-5D descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, the subject is instructed to indicate whether he or she has "no problems" (level 1), "slight problems" (level 2), "moderate problems" (level 3), "severe problems (level 4), or "extreme problems/inability" (level 5) on that day. For the EQ VAS, the participant is instructed to mark an "x" on a vertical scale at the point that best describes his or her own health on that day, where 0 represents the "worst health" he or she can imagine and 100 the "best health" he or she can imagine.
Change from Baseline in Health Utilities Index Mark 3 (HUI3) | Up to Month 24
  The HUI3 is a generic 8-item survey, which provides descriptive evidence on multiple dimensions of health status, a score for each dimension of health, and a health-related quality of life score for overall health. Health dimensions include vision, hearing, speech, ambulation/mobility, pain, dexterity, emotion and cognition. Each dimension has five or six response options. Scores on individual items are combined to given a combined health state which can then be converted to health utilities. HUI3 score ranges from 0.36 (worst) to 1 (best).
Change from Baseline in Visual Field Readings | Up to Month 24
  The progression of defects in visual fields will be assessed in both eyes using perimetry equipment.
Change from Baseline in Microperimetry Readings | Up to Month 24
  MAIA microperimetry will be conducted for both eyes to assess changes other than retinal sensitivity.
Change from Baseline in Multi-Luminance Mobility Test (MLMT) Readings | Up to Month 24
  The MLMT measures changes in functional vision, as assessed by the ability to navigate a course accurately and at a reasonable pace at different levels of environmental illumination.
Change from Baseline in Spectral Domain Optical Coherence Tomography (SD-OCT) | Up Month 24
  SD-OCT measurements will be performed after dilation of the participant's pupil.
Change from Baseline in Fundus Autofluorescence (FAF) | Up to Month 24
  Fundus Autofluorescence will be performed after dilation of the participant's pupil to assess changes in the area of viable retinal tissue.
Change from Baseline in Fundus Photography | Up to Month 24
  Seven-field colour fundus photography will be used for both eyes. Fundus photography will be performed by certified technicians following pupil dilation. Stereo photos should be performed for fields 1, 2 and 3.
Change from Baseline in Adaptive-Optics Scanning Laser Ophthalmoscopy (AO-SLO) | Up to Month 24
  Measurements will be performed after dilation of the participant's pupil.
Change from Baseline in Intraocular Pressure as Assessed by Goldmann Applanation Tonometry | Up to Month 24
  Tonometry is used to measure eye pressure. After numbing the eye with eye drop anesthesia, the Goldmann tonometer presses against the eye. The force with which the eye pushes back is used to estimate the pressure inside the eye.
Change from Baseline in Morphology of Eye as Assessed by Slit-lamp Examination | Up to Month 24
  The slit lamp exam usually forms part of a comprehensive eye exam. The participant will sit in a chair facing the slit lamp with their chin and forehead resting on a support. The doctor can use this instrument to observe the eyes in detail and determine whether or not there are any abnormalities.
Change from Baseline in Morphology of Eye as Assessed by Dilated Ophthalmoscopy | Up to Month 24
  Dilated ophthalmoscopy is performed by dilating the participant's eye to see inside the fundus of the eye and other structures using an ophthalmoscope.
Change from Baseline in Morphology of Eye as Assessed by Lens Opacities Classification System (LOCS) III Lens Grading | Up to Month 24
  LOCS III is a slit lamp based opacification grading method. Photographs of slit lamp cross-sections of the lens are used as references for grading nuclear opalescence (NO) and nuclear color (NC), and photographs of the lens seen by retroillumination are used as references for grading cortical (C) and posterior subcapsular (P) cataract. Opacification severity is graded on a decimal scale, scores can range from 0.1 to 6.9 for NO and NC and from 0.1 to 5.9 for C and P. For each opacification type the higher grading scores indicate greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (22):
- United States (10):
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Miami, Florida
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Madison, Wisconsin
- Canada (2):
  - Research Site, Montreal, Quebec
  - Research Site, Vancouver
- Research Site, Helsinki, Finland
- Research Site, Montpellier, France
- Germany (2):
  - Research Site, Bonn
  - Research Site, Tübingen
- Netherlands (2):
  - Research Site, Leiden
  - Research Site, Nijmegen
- United Kingdom (4):
  - Research Site, Leeds
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Krusenstiern L, Liu J, Liao E, Gow JA, Chen G, Ong T, Lotery AJ, Jalil A, Lam BL, MacLaren RE; XIRIUS Part 1 Study GroupXOLARIS Study Group. Changes in Retinal Sensitivity Associated With Cotoretigene Toliparvovec in X-Linked Retinitis Pigmentosa With RPGR Gene Variations. JAMA Ophthalmol. 2023 Mar 1;141(3):275-283. doi: 10.1001/jamaophthalmol.2022.6254. PMID 36757689